CLINICAL TRIAL: NCT03615170
Title: Application of Circulating Tumor DNA Test in the Diagnosis and Treatment of Patients With Advanced Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZJCH-CRC-201708
Record Dates: First submitted 2018-07-28; First posted 2018-08-03 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Rectal Neoplasms; Neoadjuvant Therapy; Circulating Tumor DNA
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Application of circulating tumor DNA detection in diagnosis and treatment of locally advanced rectal cancer. First, to explore the feasibility of ctDNA as a detection index for rectal cancer. Second, evaluate the accuracy of ctDNA detection in rectal cancer. Third, to explore whether ctDNA can be used in the evaluation of preoperative concurrent chemoradiotherapy, so as to provide guidance for subsequent treatment. Fourth, to explore the guidance value for the decision of postoperative adjuvant therapy and the frequency of reexamination. Fifth, search for possible recurrence related mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary rectal cancer；
* First treatment；
* 18 years of age or older, male or female；
* According to the indications of operation, surgical treatment can be carried out；
* According to the indications of radiotherapy, radiotherapy can be carried out；
* The physical status score of ECOG was 0~1；
* Organ function is appropriate;
* Expected survival time more than 3 months；
* During the treatment period and 6 months after treatment, contraception was not in lactation；
* The patient volunteered and signed the informed consent.

Exclusion Criteria:

* Poor compliance and failure to receive medication or follow up according to plan；
* There are other serious violations of the programme;
* At present, it has been included in other clinical trials, or at the same time, it has been included in other medical research which is judged to be incompatible with this research；
* It has a history of other cancers. Unless the cancer is completely relieved, the disease is not treated for more than 3 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced rectal cancer, who need to receive neoadjuvant radiotherapy and radical operation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 year
  Disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China